CLINICAL TRIAL: NCT03048669
Title: Continuous Quality Improvement Interventions to Improve Long Term Outcomes of Antiretroviral Therapy in Women Initiated on Therapy During Pregnancy or Breastfeeding in the Democratic Republic of Congo
Brief Title: Long Term Outcomes of Therapy in Women Initiated on Lifelong ART Because of Pregnancy in DR Congo
Acronym: CQI-PMTCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Kinshasa School of Public Health (Other)
Responsible Party: Principal Investigator, Marcel Yotebieng, Associate Professor, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2020-12018; 1R01HD087993 (NIH)
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: HIV/AIDS; Antiretroviral Therapy; Pregnancy Outcomes; HIV-exposed Infants
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The intervention will be implemented at the health facility level by the health facility staff under the supervision of health districts supervisors and investigators. As such, care providers nor investigations cannot be masked from the intervention. however, participant will not be told about the intervention or which study group they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous quality improvement (CQI) (Experimental): Quality improvement initiatives implemented at facility level using participatory data-driven approaches and on-site monitoring and supervisory support
  Interventions: Other: Continuous quality improvement
- Standard of care (No Intervention): In health districts randomized to standard of care, the same strengthening of the data collection system for the monitoring of indicators as in the intervention group will be implemented. At least once a month, a study staff will visit each clinics irrespective of their randomization to extract information for the mother-infant register into an electronic database. No report on indicators will be produced for those clinic for the duration of the study. Staff from clinics and health district bureau in the standard of care group will not be associated with the quarterly review of the indicators. The study will not influence with any other HIV service provision activity in the standard of care group.

INTERVENTIONS:
Other: Continuous quality improvement — A quality improvement team at the health district and at the clinics levels. A clinic level QI team will include at least one staff each from antenatal care (ANC), delivery/maternity, and well-child services. The head of the each QI team plus a supervisor from the health district bureau and a study team member constitute the district QI team. Immediately following randomization, we will bring together QI teams to review program and quality indicators from their clinics and across districts to identify key bottlenecks in the care delivery system and agree on an action plan to modify them. QI teams will be responsible for the implementation of the action plan at the level of their respective clinics. Every three months, using data from the monitoring system, the process will be repeated for a duration 18 months. To limit possible contamination, all staff from a randomized district/clinic who may have a dual appointment in another facility will be excluded from QI teams.
  Arms: Continuous quality improvement (CQI)

SUMMARY:
Despite the rapid adoption of the World Health Organization's 2013 guidelines, many children continue to be infected with HIV perinatally because of sub-optimal adherence to the continuum of HIV care in maternal and child health clinics (MCH). To achieve the UNAIDS goal eliminating mother-to-child HIV transmission, multiple, adaptive interventions will need to be implemented to improve adherence to the HIV continuum. The aim of this open label, parallel groups, randomized controlled trial is to evaluate the effectiveness of Continuous Quality Improvement (CQI) interventions implemented at facility and health district level to improve retention in care and virological suppression through 24 months postpartum among pregnant and breastfeeding women receiving ART in MCH clinics in Kinshasa, Democratic Republic of Congo. Prior to randomization, the current monitoring and evaluation system will be strengthen to enable collection of high quality individual patient-level data necessary for the timely production of indicators and monitoring of program outcomes to inform CQI interventions. Following randomization, in health districts randomized to CQI, quality improvement (QI) teams will be established at the district level and at MCH clinics level. For 18 months, QI teams will be brought together quarterly to identified key bottlenecks in the care delivery system using data from the monitoring system, develop an action plan to address those bottlenecks, and implement the action plan at the level of their district or clinics. If proven to be effective, CQI as designed here, could be scaled up rapidly in DRC and other resource-limited settings to accelerate progress towards the goal of an AIDS free generation.

DETAILED DESCRIPTION:
The US President's Emergency Plan for AIDS Relief (PEPFAR) goal of an AIDS-free generation, re-emphasized in PEPFAR 3.0, will not be achieved without substantial improvement in the adherence to the HIV care continuum among women in maternal and child health clinics (MCH) in resource-limited settings. In a recent meta-analysis of loss to follow-up (LTFU) across the prevention of mother-to-child transmission of HIV (PMTCT) cascade, about 50% of HIV+ pregnant women are already LTFU by delivery; within 3 months of delivery 33.9% of mother-infant pairs are also LTFU. Consequently, half of pediatric infections are currently estimated to occur in the postpartum period during breastfeeding and fewer than 40% of HEI are tested for HIV at 2-3 months. Determinants of this poor performance occur at multiple levels: healthcare delivery systems, providers, and beneficiaries (HIV-infected mothers). Current evidence suggest that beyond individual-level factors, healthcare delivery system level factors are paramount. Quality Improvement (QI) Collaborative is one of the most popular methods for organizing sustained improvement efforts at hospitals and ambulatory practices worldwide. In the Breakthrough Series approach also refer to as continuous quality improvement (CQI),10 QI teams from multiple sites across a region or country are brought together to focus on a common problem. Over one or two years, experts in clinical and performance improvement provide the group with periodic instructions and encourage the teams to share lessons learned and best practices. However, its popularity, CQI effectiveness has never been demonstrated in a randomized trial or a well-designed comparative study. The aims of the proposed study are: 1) to evaluate the effectiveness of CQI interventions in improving long-term retention in care and virological suppression in women who start lifelong ART in MCH clinics and 2) to identify modifiable health delivery system factors associated with retention in care and sustained virological suppression in women who start lifelong ART in MCH clinics. The study will be implemented in Kinshasa, Democratic Republic of Congo (DRC): an extremely resource-limited country that has struggled to emerge from decades of gross mismanagement, rampant corruption, and wars that have left its health infrastructures in shambles. We will conduct a cluster-randomized trial with health districts as the randomization unit. MCH clinics in the intervention group, will undergo CQI initiatives using participatory data-driven approaches and on-site monitoring and supervisory support. We will use surveys of health facilities, including selected staff, and service beneficiaries (HIV infected mothers) to collect data on key characteristics of the service delivery's organization and providers' and patients' perspective of the HIV care delivery performance. The main outcomes will be LTFU/retention in care, virological suppression and MTCT rates evaluated at 24 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* All women diagnosed with HIV during pregnancy or breastfeeding in the participating maternal and child health (MCH) clinics and initiated on antiretroviral therapy (ART) during the enrollment period

Exclusion Criteria:

* Refuse to participate
* Clinics will be excluded if less than 500 pregnant women (less than 5 HIV-infected pregnant women) registered for antenatal care (ANC) in the clinic in 2015

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5053 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Loss-to-follow-up | delivery, six weeks, 12 and 24 weeks postpartum
  the proportion of participants for whom the whereabouts is unknown at the evaluation time
Virological suppression | delivery, 12 and 24 months postpartum
  Proportion of participants with undetectable viral load

SECONDARY OUTCOMES:
Timely Infant HIV diagnosis | delivery, six weeks, 12 and 24 weeks postpartum
  Proportion of HIV-exposed infant with an appropriate HIV test result
Timely ART initiation | two weeks from HIV diagnosis
  Proportion of HIV-infected participants (mother or infant) initiated on ART within two weeks of diagnosis
MTCT rates | delivery, six weeks, 12 and 24 weeks postpartum
  Proportion of HIV-exposed infant who test positive for HIV
Survival | delivery, six weeks, 12 and 24 weeks postpartum
  Proportion of participating mothers and infants know to be alive

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Yotebieng, MD, PhD, Principal Investigator — Albert Einstein College of Medicine; Emile W Okitolonda, MD, PhD, Principal Investigator — Kinshasa School of Public Health
Locations (1):
- Kinshasa School of Public Health, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will include self-reported demographic and behavioral data from interviews with the subjects, clinical and laboratory data from the mother-infant pair, and blood specimens provided. Although the final dataset will be stripped of identifiers prior to release for sharing, we believe that there remains the possibility of deductive disclosure of subjects with unusual characteristics. Thus, we will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for the proposed research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed and results publish.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Yotebieng M, Mpody C, Ravelomanana NL, Tabala M, Malongo F, Kawende B, Ntangu P, Behets F, Okitolonda E; CQI-PMTCT study team. HIV viral suppression among pregnant and breastfeeding women in routine care in the Kinshasa province: a baseline evaluation of participants in CQI-PMTCT study. J Int AIDS Soc. 2019 Sep;22(9):e25376. doi: 10.1002/jia2.25376. PMID 31496051
- [Background] Yotebieng M, Behets F, Kawende B, Ravelomanana NLR, Tabala M, Okitolonda EW. Continuous quality improvement interventions to improve long-term outcomes of antiretroviral therapy in women who initiated therapy during pregnancy or breastfeeding in the Democratic Republic of Congo: design of an open-label, parallel, group randomized trial. BMC Health Serv Res. 2017 Apr 26;17(1):306. doi: 10.1186/s12913-017-2253-9. PMID 28446232
- [Background] Mpody C, Thompson P, Tabala M, Ravelomanana NLR, Malongo F, Kawende B, Behets F, Okitolonda E, Yotebieng M; CQI-PMTCT study team. Hepatitis B infection among pregnant and post-partum women living with HIV and on antiretroviral therapy in Kinshasa, DR Congo: A cross-sectional study. PLoS One. 2019 May 9;14(5):e0216293. doi: 10.1371/journal.pone.0216293. eCollection 2019. PMID 31071145
- [Background] Thompson P, Mpody C, Sayre W, Rigney C, Tabala M, Ravelomanana NLR, Malongo F, Kawende B, Behets F, Okitolonda E, Yotebieng M; CQI-PMTCT study team. Hepatitis C prevalence and quality of health services among HIV-positive mothers in the Democratic Republic of the Congo. Sci Rep. 2022 Jan 26;12(1):1384. doi: 10.1038/s41598-022-05014-3. PMID 35082320
- [Background] Zotova N, Familiar I, Kawende B, Kasindi FL, Ravelomanana N, Parcesepe AM, Adedimeji A, Lancaster KE, Kaba D, Babakazo P, Yotebieng M. HIV disclosure and depressive symptoms among pregnant women living with HIV: a cross-sectional study in the Democratic Republic of Congo. J Int AIDS Soc. 2022 Feb;25(2):e25865. doi: 10.1002/jia2.25865. PMID 35129301
- [Derived] Ndlovu KS, Pavan RR, Corry J, Gregory AC, Mahamed S, Zotova N, Tabala M, Babakazo P, Funderburg NT, Yotebieng M, Klatt NR, Kwiek JJ, Sullivan MB. The vaginal microbiome of pregnant people living with HIV on antiretroviral therapy in the Democratic Republic of Congo: a pilot study and global meta-analysis. mSphere. 2026 Jan 26:e0059725. doi: 10.1128/msphere.00597-25. Online ahead of print. PMID 41586522
- [Derived] Boisson-Walsh A, Thompson P, Fried B, Shea CM, Ngimbi P, Lumande F, Tabala M, Kashamuka MM, Babakazo P, Domino ME, Yotebieng M. Childhood immunization uptake determinants in Kinshasa, Democratic Republic of the Congo: ordered regressions to assess timely infant vaccines administered at birth and 6-weeks. Glob Health Res Policy. 2023 Dec 6;8(1):50. doi: 10.1186/s41256-023-00338-7. PMID 38057919
- See also: Continuous quality improvement interventions to improve long-term outcomes of antiretroviral therapy in women who initiated therapy during pregnancy or breastfeeding in the Democratic Republic of Congo — https://pubmed.ncbi.nlm.nih.gov/28446232/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/69/NCT03048669/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/69/NCT03048669/ICF_001.pdf